CLINICAL TRIAL: NCT00740493
Title: Eighteen Months of Oral Anticoagulant Therapy Versus Placebo After 6 Six Months of Anticoagulation for a First Episode of Idiopathic Proximal Deep Vein Thrombosis: a Multicentre Double-Blind Randomized Controlled Trial. "PADIS-TVP" Study.
Brief Title: Prolonged Anticoagulation After a First Episod of Idiopathic Proximal Deep Vein Thrombosis (PADIS TVP)
Acronym: PADIS TVP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RB06.019 PADIS TVP
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Recurrent Venous Thromboembolism; Idiopathic Deep Vein Thrombosis
Keywords: recurrent venous thromboembolism; idiopathic deep vein thrombosis; optimal duration of anticoagulation
MeSH Terms: conditions — Venous Thromboembolism | interventions — Warfarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 18 months of active warfarin therapy
  Interventions: Drug: warfarin
- 2 (Placebo Comparator): 18 months of placebo of warfarin
  Interventions: Drug: placebo of warfarin

INTERVENTIONS:
Drug: warfarin — 18 months of warfarin therapy
  Arms: 1
Drug: placebo of warfarin — 18 months of placebo of warfarin therapy
  Arms: 2

SUMMARY:
In a French multicenter double blind randomized controlled trial, the main objective is to demonstrate that, after 6 months of oral anticoagulation for a first episode of idiopathic proximal deep vein thrombosis, 18 months of warfarin therapy is associated with a lower cumulative risk of recurrent VTE and major bleeding in comparison with that on 18 months of placebo. The secondary objectives are: (1) to determine the risk of recurrent VTE after 6 months of warfarin therapy and the presence or the absence of residual lung scan perfusion defect and the persistence or not of elevated D-dimer test; and (2), to determine the impact of extended duration of anticoagulation on the risk of VTE after stopping anticoagulant therapy on a follow-up of 2 years.

DETAILED DESCRIPTION:
Rational: After 3 or 6 months of oral anticoagulation for an episode of acute venous thromboembolism (VTE), the risk of recurrent VTE is high (10 to 15% per year) in comparison with a low risk of recurrence if VTE was provoked by a major transient risk factor such as recent surgery (3% per year) independently of the initial presentation (deep vein thrombosis or pulmonary embolism). After a first episode of idiopathic VTE, 3 months of anticoagulation is associated with a very high risk of recurrence (27% per year); however, the benefit-risk of extended duration of anticoagulation (1 to 2 years) remains uncertain, mainly in relation with an increased risk of anticoagulant related bleeding. Therefore, the last ACCP conference group recommended 6 months of oral anticoagulant therapy after a first episode of idiopathic VTE. However, this recommendation is likely to be inadequate for at least two main reasons: (1) no studies compared 2 years to 6 months of anticoagulation after idiopathic VTE; and (2), if the frequency of recurrent VTE is similar after deep vein thrombosis and pulmonary embolism, however, the case fatality rate of recurrent VTE is higher after pulmonary embolism (12%) than after deep vein thrombosis (5%).

Objective : the main objective is to demonstrate that, after 6 months of oral anticoagulation for a first episode of idiopathic proximal deep vein thrombosis, 18 months of warfarin therapy is associated with a lower cumulative risk of recurrent VTE and major bleeding in comparison with that on 18 months of placebo. The secondary objectives are: (1) to determine the risk of recurrent VTE after 6 months of warfarin therapy and the presence or the absence of residual lung scan perfusion defect and the persistence or not of elevated D-dimer test; and (2), to determine the impact of extended duration of anticoagulation on the risk of VTE after stopping anticoagulant therapy on a follow-up of 2 years.

Method : French multicenter double blind randomized controlled trial. Inclusion and exclusion criteria and deep vein thrombosis diagnostic criteria have been defined. After completing 6 months of oral anticoagulation, a leg ultrasound and D-dimer testing are performed; the investigators and the patients will be unaware of the results of these tests. Then, patients are randomized to receive 18 months of warfarin therapy or 18 months of placebo (the dose of placebo will be adapted according to false computer generated INR). The investigators, the radiologists and the patients are blinded of the treatment allocation. The project has been accepted by national ethical committee and written consent will be obtained from all included patients.

Required number of patients: the expected cumulative frequency of recurrent VTE and major bleeding over 18 months is 4.5% while on warfarin therapy and 16% while on placebo. For a α risk of 5% (to falsely conclude to a true difference) and a β risk of 10% (to falsely conclude to an absence of difference), 178 patients per group should be included. As 5% of patients are expected to be loss, a total of 374 patients is required.

Feasibility: about 50 patients per year are hospitalized in our department of medicine in Brest for an acute episode of idiopathic deep vein thrombosis. Four additional centers will participate to the study and have a similar recruitment: HEGP (Pr Meyer, Dr Sanchez), CHU Antoine Béclère (Dr Parent, Pr Simmoneau), CHU Saint Etienne (Pr Mismetti, Pr Décousus), CHU Grenoble (Pr Pison, Pr Carpentier). The study will be coordinated by the Clinical Center of Investigation of Brest Hospital; "true" and "false" INR will be generated by the clinic of anticoagulant of "Ile de France" (Dr Cambus).

Clinical implications: the first consequence of the study is to demonstrate that 6 months of warfarin therapy is inadequate and should be continued for at least 18 additional months after a first episode of idiopathic proximal deep vein thrombosis. This study has also the potential to confirm or not the contribution of ultrasound of lower limb and D-dimer testing to appreciate the risk of recurrent VTE after stopping anticoagulant therapy. Lastly, the medical economical impact of such therapeutic management will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a first episode of idiopathic proximal deep vein thrombosis who have been treated during 6 months (Plus or minus 15 days) using Vitamin K antagonist with a INR between 2 and 3.

Exclusion Criteria:

* Age > 18
* warfarin hypersensibility
* unwilling or unable to give writting informed consent
* distal deep vein thrombosis or pulmonary embolism
* Proximal deep vein thrombosis which was provoked by a reversible major risk factor
* major thrombophilia (protein C, S or antithrombin deficiency, antiphospholipids antibodies, homozygous factor V Leiden)
* previous documented episode of proximale deep vein thrombosis or pulmonary embolism
* other indication for anticoagulant therapy (e.g.:atrial fibrillation, mechanic valve)
* patient on antithrombotic agent in whom antithrombotic agent should be started again after stopping anticoagulation
* pregnancy
* women without contraception
* planned major surgery in the next 18 months
* ongoing cancer or cured cancer in less than 2 years
* serious bleeding risk (e.g.: gastric ulcer)
* platelet count less than 100 Giga/l
* Life expectancy less than 18 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2007-07; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
symptomatic recurrent venous thromboembolism and serious bleedings | validated standardized objective tests

SECONDARY OUTCOMES:
mortality due to another cause than recurrent venous thromboembolism or serious bleeding | medical report and death certificates

CONTACTS AND LOCATIONS:
Overall Officials: Francis Couturaud, MD, PhD, Principal Investigator — EA3878, IFR148
Locations (14):
- France (14):
  - CHRU de Brest, Brest
  - CHU de Grenoble, Grenoble
  - Centre Hospitalier Pierre Le Damany, Lannion
  - Centre Hospitalier de Bretagne Sud, Lorient
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - AP HP Hôpital Hôtel Dieu, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - CHU de POITIERS, Poitiers
  - Centre Hospitalier de Cornouaille, Quimper
  - CHU de Rennes, Rennes
  - Centre Hospitalier de Saint Brieuc, Saint-Brieuc
  - Hôpital de Rangueil, Toulouse
  - CHU de Tours, Tours
  - Centre Hospitalier Intercommunal, Vernon

REFERENCES:
- [Derived] Couturaud F, Pernod G, Presles E, Duhamel E, Jego P, Provost K, Pan-Petesch B, Sollier CBD, Tromeur C, Hoffmann C, Bressollette L, Lorillon P, Girard P, Le Moigne E, Le Hir A, Guegan M, Laporte S, Mismetti P, Lacut K, Bosson JL, Bertoletti L, Sanchez O, Meyer G, Leroyer C, Mottier D; "PADIS-DVT" investigators. Six months versus two years of oral anticoagulation after a first episode of unprovoked deep-vein thrombosis. The PADIS-DVT randomized clinical trial. Haematologica. 2019 Jul;104(7):1493-1501. doi: 10.3324/haematol.2018.210971. Epub 2019 Jan 3. PMID 30606789